CLINICAL TRIAL: NCT00383968
Title: Prevalence of Chronic KIdney Disease in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Other Study IDs: 06GS009CHS
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Last update posted 2006-10-04 (Estimated); Status verified 2006-10

CONDITIONS: Hypertension; Chronic Kidney Disease
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Prevention of progressive renal disease needs a clear understanding of prevalence of early stage of chronic kidney disease in a community. Even in developed countries most subjects in early stages of chronic kidney disease go largely undiagnosed and untreated. Targeted screening could identify a greater numbers of individuals at risk then a general public screening (11). It is economically more feasible to perform in a country like Pakistan. Hypertension and diabetes are highly prevalent in South-Asia.It is anticipated that if target screening of hypertensive population is performed especially of an age group in which intervention might be expected to have maximal benefit it will not only help to identify from a large number of patients with essential hypertension destined to develop or in the course of advancing towards end stage renal disease but will also unearth mislabeled "essential hypertension" that have underlying primary renal disease. This later group may belong to socio-economic disadvantaged population who have limited access to health care and have never been investigated properly. The aim of the Study is to detect sub-clinical chronic kidney disease in hypertensive patients at community level and to identify associated risk factors.

DETAILED DESCRIPTION:
This will be Cross sectional or prevalent study targeting diagnosed hypertensives aged 40 and above years, in middle to low socio-economic settings of Karachi. This proposed study will be nested in the existing Wellcome Trust funded study. The parent study is designed to determine the impact of a unique community versus high risk approach to control BP in Karachi, Pakistan In that ongoing Factorial design, individuals aged ≥40 who are found hypertensive in the 12 clusters (each containing 250 households) are being randomized to different interventions for their BP control. All participants enrolled in that study had urine examination for proteinuria and serum creatinine measurements at baseline to assess their renal status. For the proposed study the identified hypertensive (from parent study) who had either shown proteinuria and or had elevated serum creatinine (more then 1.2 for females and 1.4 mg/dl for males) at baseline will be approached. Serum creatinine levels exceeding above mentioned cut-off levels, are only reached when GFR is<60ml/min/m². As mentioned above in order to classify these subjects as having chronic kidney disease these abnormalities must be demonstrated to persist for at least three months. A repeat serum creatinine measurement and urine examination for proteinuria will be performed in the present study, by obtaining blood sample and urine sample respectively from these subjects. As a period of three months have already passed since the baseline investigations were done, all subjects who will show persistent abnormalities in either or both test will fall into chronic kidney disease group. The repeated testing to confirm presence of CKD will include, measurement of serum creatinine and urinary albumin/creatinine ratio (>30mg/g) in an untimed urine specimen. This method has been recommended as the preferred screening strategy. A set questionnaire will be filled by interviewing the patient and risk factors for the presence of renal disease will be analyzed based on this information.

The data collection will be done through structured questionnaire and diagnosis will be made on the basis of their persistently elevated kidney biomarkers.

ELIGIBILITY:
Inclusion criteria:

* Known hypertensives aged 40 and above with microalbuminuria and/or elevated serum creatinine on first evaluation.
* Hypertension: Systolic blood pressure ≥140, and /or diastolic blood pressure ≥ 90 with or without antihypertensive drugs.
* Microalbuminuria:

  * Albumin concentration of 20-200mg/L, with albumin-to-creatinine ratio of 3-30mg/mmol or 30-300mg/g
  * Female: 3.0-30.0mg/mmol or 30-300mg/g
  * Male: 2.0-20.0mg/mmol or 20
* Elevated Serum creatinine:

  * Female: >1.2mg/dl
  * Male: >1.4mg/dl

Exclusion Criteria:

* Known diabetics will be excluded.
* unable to give informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248
Dates: Start 2006-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Study Director — Aga Khan University; Muslima A Ejaz, MBBS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan